CLINICAL TRIAL: NCT00167635
Title: Nursing Management of Irritable Bowel Syndrome: Improving Outcomes
Brief Title: Nursing Management of Irritable Bowel Syndrome:Improving Outcomes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Margaret Heitkember, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12707-C; 2R01NR04142-5; 97-3895-C 11; 2R01NR004142 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Cognitive-behavioral intervention; Psychological distress; Quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Face-to-Face Individualized Comprehensive Self-Management (CSM-FF) Group. Participants in the individualized CSM-FF group will be scheduled for 9 weekly sessions with the nurse therapist followed by post-intervention follow-up assessment.
  Interventions: Behavioral: cognitive-behavioral
- 2 (Experimental): Telephone Individualized Comprehensive Self-Management (CSM-TEL) Group. Participants in the individualized CSM-FTF group will initially have 2 face-to-face meetings with the nurse therapist, 6 sessions over the phone and the final session face-to-face at 9 weeks.
  Interventions: Behavioral: cognitive-behavioral
- 3 (No Intervention): Usual Care Control Group (UC). Following randomization the participants in the control group will receive two short phone calls to maintain contact during the comparable 9-week intervention in the treatment groups.
  Interventions: Behavioral: cognitive-behavioral

INTERVENTIONS:
Behavioral: cognitive-behavioral — Cognitive-behavioral over 9 weeks
  Other Names: Usual care

SUMMARY:
The purpose of this study is 1) to determine whether a comprehensive self-management intervention is effective in a sample that includes men and women with irritable bowel syndrome, and 2) to determine whether the comprehensive self-management intervention is as effective when delivered over the telephone as compared to a face-to-face approach.

DETAILED DESCRIPTION:
Randomization and Intervention Phase. Upon completing the baseline assessment phase, participants will be randomized to one of 3 treatment groups. A customized computer program will be used to do the randomization in an adaptive manner that ensures the 3 groups remain fairly balanced with respect to possible important predictors of outcomes: age, sex, predominant stool pattern (alternating, constipation-predominant or diarrhea-predominant), and severity of IBS symptoms and psychological symptoms at baseline. When each new participant is randomized, the program will adjust the probabilities of assignment to the three groups so that there is a higher probability of assignment to the group that results in the best balance.

Intervention Groups. Face-to-Face Individualized Comprehensive Self-Management (CSM-FF) Group. Participants in the individualized CSM-FF group will be scheduled for 9 weekly sessions with the nurse therapist followed by post-intervention follow-up assessment.

Telephone Individualized Comprehensive Self-Management (CSM-TEL) Group. Participants in the individualized CSM-TEL group will initially have 2 face-to-face meetings with the nurse therapist, 6 sessions over the phone and the final session face-to-face at 9 weeks.

Usual Care Control Group (UC). Following randomization the participants in the control group will no receive any contacts during the comparable 9-week intervention in the treatment groups.

Follow-up Phase. Participants in all 3 groups will be reassessed at 3-mo, 6-mo, and 12-mo post randomization. At this time the participants will complete questionnaires, a 4 week diary and collect 4 urines.

ELIGIBILITY:
Inclusion Criteria:

* Irritable Bowel Syndrome

Exclusion Criteria:

* GI pathology (organic disease)
* Co-morbid pain disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2003-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | baseline, and 3 months, 6 months, 12 months post randomization
Psychological distress | baseline, and 3 months, 6 months, 12 months post randomization
Cognitive Scale for Functional Bowel Disorders (CFBD) describes 25 cognitive beliefs related to functional bowel disorders. | baseline, and 3 months, 6 months, 12 months post randomization
Health Related Quality Of Life (HRQOL) will be measures with the Disease Specific Questionnaire-IBS (IBS-DSQ), a 42-item questionnaire. | baseline, and 3 months, 6 months, 12 months post randomization

SECONDARY OUTCOMES:
Sleep disturbance | baseline, and 3 months, 6 months, 12 months post randomization
Sexual dysfunction | baseline, and 3 months, 6 months, 12 months post randomization
Catecholamine and cortisol levels (urine) | baseline, and 3 months, 6 months, 12 months post randomization
Stool frequency/consistency | baseline, and 3 months, 6 months, 12 months post randomization
Health care utilization | baseline, and 3 months, 6 months, 12 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M Heitkemper, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Northgate Executive 1, Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Heitkemper MM, Jarrett ME, Levy RL, Cain KC, Burr RL, Feld A, Barney P, Weisman P. Self-management for women with irritable bowel syndrome. Clin Gastroenterol Hepatol. 2004 Jul;2(7):585-96. doi: 10.1016/s1542-3565(04)00242-3. PMID 15224283
- [Derived] Yang PL, Burr RL, Buchanan DT, Pike KC, Kamp KJ, Heitkemper MM. Indirect effect of sleep on abdominal pain through daytime dysfunction in adults with irritable bowel syndrome. J Clin Sleep Med. 2020 Oct 15;16(10):1701-1710. doi: 10.5664/jcsm.8658. PMID 32620184
- [Derived] Kamp KJ, Weaver KR, Sherwin LB, Barney P, Hwang SK, Yang PL, Burr RL, Cain KC, Heitkemper MM. Effects of a comprehensive self-management intervention on extraintestinal symptoms among patients with IBS. J Psychosom Res. 2019 Nov;126:109821. doi: 10.1016/j.jpsychores.2019.109821. Epub 2019 Aug 29. PMID 31499231
- [Derived] Han CJ, Kohen R, Jun S, Jarrett ME, Cain KC, Burr R, Heitkemper MM. COMT Val158Met Polymorphism and Symptom Improvement Following a Cognitively Focused Intervention for Irritable Bowel Syndrome. Nurs Res. 2017 Mar/Apr;66(2):75-84. doi: 10.1097/NNR.0000000000000199. PMID 28252569